CLINICAL TRIAL: NCT06862440
Title: Detection of Fertile Window and Ovulation with At-Home Kegg Fertility Monitor: a Comparative Study with Standardized Cervical Mucus Observations and Urine Hormone Measurements
Brief Title: Kegg Fertility Study
Acronym: CMTrak-US
Status: Recruiting | Type: Observational
Sponsor: Lady Technologies Inc (Industry)
Responsible Party: Principal Investigator, Jan Rydfords, Principal Investigator, Lady Technologies Inc
Other Study IDs: LT-002
Record Dates: First submitted 2025-01-23; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Fertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Kegg Cohort: Daily data collection of kegg electrical impedance, urine hormone test, and basal body temperature on non-bleeding days. Data will be collected for 3 cycles.
  Interventions: Device: Kegg

INTERVENTIONS:
Device: Kegg — Fertility status monitor

SUMMARY:
Fertility Awareness Based Methods (FABMs), such as calendar tracking, basal body temperature (BBT), and monitoring cervical mucus, are widely used but may have limitations in accurately detecting the complete fertility window. Serum hormone measurements and transvaginal ultrasound are more accurate at determining time of ovulation and fertile window, but are costly and inconvenient. Urine-based luteinizing hormone (LH) tests offer improvement. However, LH surge typically occurs 24 to 36 hours prior to ovulation, only capturing the later portion of the fertile window.

A novel approach involves using electrical impedance to track compositional changes in cervical mucus, providing real-time, at-home data. The Kegg device (Lady Technologies Inc, San Francisco, CA, USA) is an intravaginal device that measures cervical mucus impedance to monitor fertility status. Previous studies show it has higher sensitivity, specificity, and accuracy compared to BBT alone in determining the ovulation window. This method offers a cost-effective and practical alternative for at-home fertility tracking.

The objectives of this study are to:

1. evaluate the association between Kegg electrical impedance readings and cervical mucus observations with regard to determining fertility status; and
2. compare the accuracy of Kegg electrical impedance readings with hormone urine strips in identifying the complete fertile window determined by cervical mucus observations.

ELIGIBILITY:
Inclusion Criteria:

1. Biological female
2. Age between 18-40 years old
3. Participant has provided signed informed consent
4. Completed cervical mucus observation training
5. Owns and uses daily a smart device meeting the following requirement: Apple iPad or iPhone running iOS 13 or newer, or Apple Watch running WatchOS 6.0 or newer, or Android operating system of 6.0 or newer
6. Has readily accessible internet
7. Legal residents of the continental United States, excluding Alaska and Hawaii.

Exclusion Criteria:

1. Participant is unable to read and understand English
2. Postmenopausal women
3. Women with hysterectomy
4. Pregnancy
5. Hormonal or intrauterine contraceptives or other hormone use prior to start of study enrollment [No oral hormonal contraceptives or other hormones for at least one month, no implantable contraceptives or hormonal or non-hormonal intrauterine device for at least two months (~2 cycles), no injectable hormonal contraceptives or other hormones in past 9 months from the most recent injection and resumption of regular menstrual cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Mucus characteristics quantified by electrical impedance readings | Daily on non-bleeding days for 3 cycles (each cycle is approximately 28 days)
  Electrical impedance measured daily on non-bleeding days for 3 menstrual cycles.
Cervical mucus scores | Daily on non-bleeding days for 3 cycles (each cycle is approximately 28 days)
  Participant self-graded scores of cervical mucus appearance using standardized scoring system
Urine hormone test results | Daily on non-bleeding days for 3 cycles (each cycle is approximately 28 days)
  Hormone changes in E1G (estrogen), LH, luteinizing hormone, and PdG (progesterone) measured by urine hormone test

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Technologies Inc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tabbaa S, Hambright S, Sikes KJ, Levy G, Rydfors J. The effectiveness of cervical mucus electrical impedance compared to basal body temperature to determine fertility window. Contracept Reprod Med. 2024 May 6;9(1):20. doi: 10.1186/s40834-024-00276-w. PMID 38705979